CLINICAL TRIAL: NCT00515905
Title: Lung: One-lung Ventilation: Expression of Pulmonary Inflammatory Mediators After Deflation and Re-expansion of the Lung During Thoracic Surgery
Brief Title: One-lung Ventilation: Expression of Pulmonary Inflammatory Mediators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Beatrice Beck-Schimmer, University of Zurich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: StV 20-2004
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Last update posted 2010-09-15 (Estimated); Status verified 2008-03

CONDITIONS: Thoracic Surgery With One-lung Ventilation
MeSH Terms: interventions — Sevoflurane; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sevoflurane/propofol — Sevoflurane/propofol

SUMMARY:
One-lung ventilation; organ protection; volatile anesthetics

One-lung ventilation has become a common procedure for thoracoscopic surgery. Two hypothesis will be tested in this study:

1. Are inflammatory mediators increased in the re-ventilated lung after short-period pulmonary collapse?
2. Does Sevoflurane influence the production of inflammatory mediators in the re-inflated lung? Therefore, this study will elucidate the potential protective effect of a volatile anaesthetic (sevoflurane) on the production of inflammatory mediators by the respiratory compartment of the lung, i.e. the alveolar epithelium.

   * Trial with immunomodulatory product / biological

ELIGIBILITY:
Inclusion criteria:

* Thoracic surgery (thoracotomy, thoracoscopy) with one-lung ventilation

Exclusion criteria:

* Immunosuppressive therapy
* Ongoing inflammatory processes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2004-10; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
One-lung ventilation measurement in the re-ventilated lung after short-period pulmonary collapse | Sep 07

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- University Hospital of Zurich, Zurich, Switzerland